CLINICAL TRIAL: NCT04193072
Title: Assessment of Imagery Ability in Children With Obstetric Brachial Plexus Palsy
Brief Title: Imagery Ability in Obstetric Brachial Plexus Palsy
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Nursena Şengün, Physiotherapist, Istanbul Medipol University Hospital
Other Study IDs: 10840098-604.01.01-E.10507
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Brachial Plexus Palsy; Image, Body
Keywords: brachial plexus; imagery; body image; sensation; questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obstetric brachial plexus palsy
  Interventions: Behavioral: Assessment of imagery ability
- Healthy
  Interventions: Behavioral: Assessment of imagery ability

INTERVENTIONS:
Behavioral: Assessment of imagery ability — Movement imagery, kinesthetic imagery, and visual imagery ability assessed.

SUMMARY:
Obstetric brachial plexus palsy (OBPP) is the paralysis of the ipsilateral upper extremity after a brachial plexus injury that occurs during labor. Imagery is to rehearse sensorial experiences in the mind such as auditory, visual, tactile, olfactory, gustatory or kinesthetic sensation. Imagery is used as a new technique in rehabilitation recently. Various studies have reported the importance of imagery and using imagery as a rehabilitation technique in different neurologic and orthopedic conditions. This study aimed to evaluate imagery ability in children with OBPP.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 8-18 years
* Children with OBPP Narakas's classification system rating of Type 1, Type 2a, Type 2b, or Type 3
* Standardized mini-mental state examination score >24
* With no physical or neurological condition affecting motor development

Exclusion Criteria:

* Narakas's classification system rating of Type 4
* Standardized mini-mental state examination score <24
* Surgical operation in last 6 months
* Physical or neurological conditions
* Refuse to attend to the study

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with obstetric brachial plexus palsy and healthy children.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-01-27 (Actual); Study Completion 2018-03-25 (Actual)

PRIMARY OUTCOMES:
Movement Imagery Questionnaire-3 | 2 weeks
  Movement Imagery Questionnaire-3 is a 12-item questionnaire to assess an individual's ability to achieve specific four movements using internal visual imagery, external visual imagery, and kinesthetic imagery.
Kinesthetic and Visual Imagery Questionnaire-20 | 2 weeks
  Kinesthetic and Visual Imagery Questionnaire-20 assess an individual's ability to visualize and feel imagined movements.
Active Movement Scale | 1 week
  Active Movement Scale evaluates 15 joint movements in the upper extremity against gravity and gravity-eliminated positions. Each movement is given a score between 0-7: 0 means no contraction, 7 means full range of motion.
Narakas's Sensory Grading System | 1 week
  Narakas's Sensory Grading System evaluates the response to painful stimuli in the upper extremity with 0-3-point scale: 0 indicates no reaction, 3 indicates a normal reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Nursena Şengün, PT, MSc, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided